CLINICAL TRIAL: NCT02657265
Title: Prospective Multicenter Randomized Study Comparing Two Standard Treatments: SpineJack® System and Conservative Orthopedic Management in Acute Traumatic Vertebral Fractures Types A1 and A3.1 According to the Magerl Classification
Brief Title: SpineJack® Versus Conservative Treatment Study (SPICO Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vexim SA (Industry)
Collaborators: Statitec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EU2014-09
Record Dates: First submitted 2016-01-05; First posted 2016-01-15 (Estimated); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Spinal Fractures; Vertebral Compression Fractures; Back Injuries; Trauma
MeSH Terms: conditions — Spinal Fractures; Back Injuries; Wounds and Injuries | interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SpineJack® system (Experimental): Spine fracture management
  Interventions: Device: SpineJack system
- Conservative management (Active Comparator): Surgical corset according to measurement's impression, rigid corset with sternal support
  Interventions: Device: Conservative management

INTERVENTIONS:
Device: SpineJack system — Spine fracture management for traumatic vertebral compression fracture
  Arms: SpineJack® system
Device: Conservative management — Surgical corset according to measurement's impression, rigid corset with sternal support
  Arms: Conservative management

SUMMARY:
This study will compare two standard treatments in acute stable traumatic vertebral fractures (types A1 and A3.1 by Magerl Classification). The two treatments are as follows:

1. SpineJack® system
2. Conservative Orthopedic Management consisting of brace and pain medication.

DETAILED DESCRIPTION:
100 subjects (18 to 60 years old) will be enrolled (1:1) with one to two painful traumatic fractures, non-pathological (types A1 and A3.1 by Magerl Classification).

Subjects will be followed at admission, procedure, discharge, 1 month, 3 months, 12 months and 24 months post Vertebral Compression Fracture (VCF) reduction procedure or the set-up of the brace.

The estimated enrollment period is 12 months and each patient should perform a 24 months follow-up period. Therefore, the total study duration is estimated to be 36 months for the complete study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed the consent form
2. Male or Female between 18 and 60 years old
3. One to two painful traumatic fractures, non-pathological, traumatic vertebral fracture is less than 10 days, between T11 and L5, type A1 and A3.1 according to Magerl classification. All the fractures should meet the inclusion criteria (deformity, etiology, technical possibility of performing the procedure).
4. Vertebral kyphosis angle >10°
5. Patient is eligible to treatment with brace
6. Technical feasibility of a SpineJack® procedure and brace 1 to 5 days after screening/baseline

Exclusion Criteria:

1. Vertebral fracture more than 10 days old
2. Spontaneous osteoporotic vertebral fracture
3. Neurological signs or symptoms related to the vertebral fracture
4. Vertebral kyphosis angle >30°
5. Active systemic or local infection at baseline
6. Patient with substance abuse
7. History of intolerance or allergic reaction to titanium or acrylic compounds
8. Fracture geometry making the insertion of the implant impossible
9. Malignant lesions
10. Any other medical illness or condition that, in the investigator's opinion, is likely to impair long-term follow-up (e.g., cancer) or greatly increase the risk of surgery*
11. Patient on long-term steroid therapy (steroid dose ≥ 30 mg /day for > 3 months)
12. Patient presenting with a non-correctable spontaneous or therapeutic coagulation disorder.
13. Non-compliant patient: Impossibility to participate in the study and to be followed-up for 2 years.
14. Participating in any other investigational study
15. Female patients who are pregnant, breastfeeding, or planning to get pregnant during the course of the study
16. Patient not affiliated to social security *: including but not limited to patients with contraindications for general anesthesia (surgeon expertise)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2020-05-25 (Actual)

PRIMARY OUTCOMES:
VAS | 1 and 12 months follow-up
  Mean Visual Analogue Scale (VAS) back pain score at 1 and 12 months follow-up

SECONDARY OUTCOMES:
Oswestry Disability Index | Screening/baseline, immediat post-op, 1, 3, 12 and 24 months
EQ-5D | Screening/baseline, immediat post-op, 1, 3, 12 and 24 months
Kyphotic angle | Screening/baseline, immediat post-op, 1, 3, 12 and 24 months
Regional Kyphotic Angle | Screening/baseline, immediat post-op, 1, 3, 12 and 24 months
Evaluation of safety through evaluation of adverse events | Screening/baseline, immediat post-op, 1, 3, 12 and 24 months
Costs comparison of overall treatments | Screening/baseline, immediat post-op, 1, 3, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Vital, Prof., Principal Investigator — Hopital Pellegrin - Bordeaux
Locations (9):
- France (9):
  - Hopital Jean Minjoz Besancon, Besançon
  - CHU de Bordeaux - Hopital Pellegrin, Bordeaux
  - CHU Brest, Brest
  - Centre Hospitalier De Chambéry, Chambéry
  - CHU de Dijon, Dijon
  - APHM, Hopital Nord Marseille, Marseille
  - CHU de Rennes, Rennes
  - CHU de Rouen-Hopital Charles Nicolle, Rouen
  - Centre Hospitalier Privé Saint Grégoire, Saint-Grégoire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ould-Slimane M, Petit A, Gille O, Kaya JM, Touta A, Lebhar J, Grelat M. A prospective multicenter randomized study comparing the SpineJack system and nonsurgical management with a brace in acute traumatic vertebral fractures: the SPICO study. J Neurosurg Spine. 2024 Mar 1;40(6):790-800. doi: 10.3171/2023.12.SPINE23824. Print 2024 Jun 1. PMID 38427996